CLINICAL TRIAL: NCT04898985
Title: The Leukemia and Lymphoma Society (LLS) T-cells in Blood Cancer and COVID-19
Acronym: LLST-Cells
Status: Suspended | Type: Observational
Why Stopped: Recruitment was completed for initial evaluation of T-cell response to early Covid-19
Sponsor: Larry Saltzman, MD (Other)
Responsible Party: Sponsor-Investigator, Larry Saltzman, MD, Principal Investigator, Blood Cancer United
Organization: Blood Cancer United (Other)
Other Study IDs: LLSC19-002
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 500 patients in the LLS COVID-19 Registry with no/limited antibody response: Five hundred (500) patients participating in the LLS COVID-19 Registry, who have shown either no antibody or limited antibody response by way of the Spike Antibody test to one of the vaccinations authorized for emergency use (EUA) by FDA will participate in this Research Study.
  Interventions: Diagnostic Test: ImmunoSEQ
- 500 patients also participating in the LLS COVID-19 Registry with antibody response: 500 patients with similar blood cancer diagnosis, also participating in the LLS COVID-19 Registry, who have shown full Spike antibody response to one of the vaccinations authorized for emergency use (EUA) by FDA will also be enrolled in this Research Study for comparison (as a control arm) and will also be followed for at least 10 years (in the COVID-19 Registry).
  Interventions: Diagnostic Test: ImmunoSEQ

INTERVENTIONS:
Diagnostic Test: ImmunoSEQ — experiment assay

SUMMARY:
Five hundred (500) patients participating in the LLS COVID-19 Registry, who have shown either no antibody or limited antibody response by way of the Spike Antibody test to one of the vaccinations authorized for emergency use (EUA) by FDA will participate in the LLS T-cells, Blood Cancer and COVID-19 Clinical Research Study. They will be followed for at least ten years (in the COVID-19 Registry). In addition, 500 patients with similar blood cancer diagnosis, also participating in the LLS COVID-19 Registry, who have shown full Spike antibody response to one of the vaccinations authorized for emergency use (EUA) by FDA will also be enrolled the LLS T-cells, Blood Cancer and COVID-19 Clinical Research Study for comparison (as a control arm) and will also be followed for at least 10 years (in the COVID-19 Registry).

DETAILED DESCRIPTION:
LLS has partnered with Adaptive Biotechnologies, to provide their ImmunoSEQ research assay to accumulate data about patients with blood cancer, who have received an FDA authorized vaccination, and depending on the type of cancer, have developed no antibodies or limited antibodies, to determine if these individuals have developed T-cells. While antibodies have been a mainstay in measuring the immune response to vaccines, for COVID-19, it has become clear that the T-cell response is necessary for a complete picture of immunity.

Five hundred (500) patients participating in the LLS COVID-19 Registry, who have shown either no antibody or limited antibody response by way of the Spike Antibody test to one of the vaccinations authorized for emergency use (EUA) by FDA will participate in this Research Study. They will be followed for at least ten years (in the COVID-19 Registry). In addition, 500 patients with similar blood cancer diagnosis, also participating in the LLS COVID-19 Registry, who have shown full Spike antibody response to one of the vaccinations authorized for emergency use (EUA) by FDA will also be enrolled in this Research Study for comparison (as a control arm) and will also be followed for at least 10 years (in the COVID-19 Registry).

Patients will be advised that ImmunoSEQ is not an FDA authorized/approved diagnostic assay and that as a "research assay" results cannot be shared with them.

The process for patients to participate in the LLS T-cells, Blood Cancer and COVID-19 Clinical Research Study includes:

* LLS will identify who is eligible and who will be invited to participate in this study.
* Ciitizen will send an email to eligible patients to invite them to participate.
* Patients will be sent a study page Password and instructed not to share it.
* Eligible patients will visit the LLS T-cells, Blood Cancer and COVID-19 Clinical Research Study-specific page. Patients will be advised to read the entire Consent Form and, if satisfied, patients will be asked to enter the password and then sign the pop-up consent by entering Name, Email, and Phone Number.
* Within 24 hours, patients will receive an email notifying them that their unique lab slip has been uploaded into their Ciitizen account. To access, patients will login to their Ciitzen account with their User ID/Password credentials for the LLS T-cells, Blood Cancer and COVID-19 Clinical Research Study.
* Patients will schedule a blood draw at a LabCorp facility.
* Note: Patients will be informed that Study results CAN NOT be shared with patients individually; only in aggregate once the Study concludes.
* And, at any time, should patients have any questions, LLS contact information is on the front page of the Informed Consent document.

After providing electronic signature to the informed consent, this Research Study requires patients who have received an FDA authorized vaccination, and depending on the type of cancer, have developed no antibodies or limited antibodies, to provide one blood sample of less than 3ccs drawn at any LabCorp facility (at no cost to patients). LabCorp facility locations can be found online at https://www.labcorp.com/labs-and-appointments-advanced-search.

ELIGIBILITY:
Inclusion Criteria:

* Select patients participating in the LLS COVID-19 Registry will be invited to enroll

Exclusion Criteria:

* People who have not participated in the LLS COVID-19 Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Five hundred (500) patients participating in the LLS COVID-19 Registry, who have shown either no antibody or limited antibody response by way of the Spike Antibody test to one of the vaccinations authorized for emergency use (EUA) by FDA will participate in this Research Study.
  500 patients with similar blood cancer diagnosis, also participating in the LLS COVID-19 Registry, who have shown full Spike antibody response to one of the vaccinations authorized for emergency use (EUA) by FDA will also be enrolled in this Research Study for comparison (as a control arm) and will also be followed for at least 10 years (in the COVID-19 Registry).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2031-05-20 (Estimated); Study Completion 2031-05-20 (Estimated)

PRIMARY OUTCOMES:
Number of people who have developed T cells from a COVID-19 vaccination | 2 years
  ImmunoSEQ research assay to accumulate data about patients with blood cancer, who have received an FDA authorized vaccination, and depending on the type of cancer, have developed no antibodies or limited antibodies, to determine if these individuals have developed T-cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Lymphoma and Leukemia Society, Rye Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No
Patients will be advised that ImmunoSEQ is not an FDA authorized/approved diagnostic assay and that as a "research assay" results cannot be shared with them.